CLINICAL TRIAL: NCT01250561
Title: Reduction of Postherpetic Neuralgia in Herpes Zoster
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Clinical Studies, Texas (Other)
Responsible Party: Stephen Tyring, Center for Clinical Studies
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCS-06-001
Record Dates: First submitted 2010-11-29; First posted 2010-12-01 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Herpes Zoster; Post-herpetic Neuralgia
Keywords: gabapentin; valacyclovir; phn; shingles
MeSH Terms: conditions — Herpes Zoster; Neuralgia, Postherpetic | interventions — Gabapentin; Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Gabapentin — gabapentin 300mg/day, titrated up weekly to max tolerated dose or 3600mg/day (whichever is lower), for 4-9 weeks
Drug: Valacyclovir — valacyclovir 1000mg three-times daily x 7 days

SUMMARY:
The addition of gabapentin therapy to standard antiviral treatment with valacyclovir in acute herpes zoster patients will decrease the incidence of post-herpetic neuralgia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of 50 years of age and older.
* Patients with a clinical diagnosis of uncomplicated herpes zoster presenting within the first 72 hours of vesicles.
* Patients who are willing and able to comply with the requirements of the study.
* Patients who are willing and able to give written informed consent.
* Average pain score pre-therapy greater or equal than 4 on 10-point Likert scale.

Exclusion Criteria:

* Sexually-active women of childbearing potential, including postmenopausal women less than 1 year since last menses, not employing adequate contraception (approved oral contraceptive, intrauterine device, barrier methods or total abstinence).
* Pregnant females and nursing mothers.
* Patients with immune dysfunction including congenital immune deficiency, active malignancy of any type, collagen vascular diseases, organ or bone marrow transplantations, known infection with HIV or severe atopic dermatitis.
* Patients who have received cytotoxic drugs or immunosuppressive therapy (e.g., chronic systemic corticosteroids) within the previous 3 months.
* Patients with evidence of cutaneous or visceral dissemination of herpes zoster infection (cutaneous dissemination is defined as > 20 discrete lesions outside adjacent dermatomes).
* Patients who have received systemic anti-VZV medications or immunomodulatory medications (including interferon) within the previous 4 weeks.
* Patients currently receiving probenecid.
* Patients with impaired renal function: calculated creatinine clearance of <30 mL/min using Cockcroft and Gault formula.
* Patients with abnormal liver function (alanine transaminase (ALT) or aspartate;transaminase (AST) levels greater than five times the upper limit of the normal range).
* Patients with a history of intolerance or hypersensitivity to acyclovir, penciclovir, valacyclovir, famciclovir or gabapentin.
* Patients currently receiving therapy with gabapentin or tricyclic antidepressants.
* Patients with clinical evidence of ocular involvement of herpes zoster. Patients with herpes zoster of the ophthalmic branch of the trigeminal nerve without evidence of ocular involvement will be included.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2002-02; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with zoster pain at 6 months

SECONDARY OUTCOMES:
Proportion of patients with zoster pain at 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Tyring, MD, PhD, Principal Investigator — Center for Clinical Studies
Locations (1):
- Center for Clinical Studies, Houston, Texas, United States

REFERENCES:
- [Derived] Lapolla W, Digiorgio C, Haitz K, Magel G, Mendoza N, Grady J, Lu W, Tyring S. Incidence of postherpetic neuralgia after combination treatment with gabapentin and valacyclovir in patients with acute herpes zoster: open-label study. Arch Dermatol. 2011 Aug;147(8):901-7. doi: 10.1001/archdermatol.2011.81. Epub 2011 Apr 11. PMID 21482862